CLINICAL TRIAL: NCT07038018
Title: External Validation of Artificial Intelligence-Enabled Electrocardiograms for the Detection of Reduced Left Ventricular Ejection Fraction
Brief Title: External Validation of Artificial Intelligence-enabled Electrocardiography (AI-ECG) for the Detection of Left Ventricular Dysfunction (LVD)
Status: Not yet recruiting | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wei-Ting Liu, Clinical Doctor, Principal Investigator, Tri-Service General Hospital
Other Study IDs: B202405084
Record Dates: First submitted 2025-06-16; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Disease
Keywords: left ventricular dysfunction; artificial intelligence
MeSH Terms: conditions — Heart Diseases; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AI-ECG Algorithm — AI-ECG Algorithm to detect LVEF<=40%

SUMMARY:
This is a multi-center, retrospective study evaluating the performance of an artificial intelligence-enabled electrocardiography (AI-ECG) algorithm in detecting reduced left ventricular ejection fraction (LVEF ≤ 40%). All included patients from participating hospitals must have undergone a digital 12-lead electrocardiogram (ECG) and an echocardiogram with assessment of LVEF within seven days. The AI-ECG algorithm will be applied to evaluate its diagnostic performance, which will be further assessed across subgroups stratified by demographic characteristics and clinical factors.

DETAILED DESCRIPTION:
Data were collected from 13 hospitals, excluding the medical center that developed the artificial intelligence-enabled electrocardiography (AI-ECG) algorithm. The primary objective of the study was to evaluate the sensitivity and specificity of the AI-ECG model in detecting left ventricular dysfunction, defined as left ventricular ejection fraction (LVEF) ≤ 40%. To ensure clinical applicability, predefined thresholds required both sensitivity and specificity to exceed 0.80 in external validation cohorts. Sample size calculations were based on testing the null hypothesis that sensitivity equals 0.80. In the development hospital cohort, the model demonstrated a sensitivity of 0.869 and a specificity of 0.896. With a two-sided significance level (α) of 0.05 and a power of 90%, an estimated 310 cases of LVEF ≤ 40% were required.

Given that the prevalence of left ventricular dysfunction was 4% in the development hospital cohort but expected to be lower-between 2.5% and 3%-in external validation settings (i.e., regional and local hospitals), the total sample size needed to accrue the target number of cases was estimated to range between 10,333 and 12,400 patients. To achieve this, six regional hospitals and seven local hospitals were selected as external validation sites. Because both electrocardiography and echocardiography were required within a seven-day interval-leading to anticipated exclusions-approximately 1,500 patients were targeted from each regional hospital and 500 from each local hospital, resulting in a final target sample size of approximately 12,500 patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with ECGs and an echocardiogram within 7 days

Exclusion Criteria:

* Missing ECG signals
* Missing LVEF assessment in echocardiograms

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with ECGs and an echocardiogram within 7 days
Sampling Method: Probability Sample
Enrollment: 12500 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The Sensitivity and specificity of AI-ECG model for left ventricular ejection fraction ≤ 40% | within 7 days
  The primary objective of the study was to evaluate the sensitivity and specificity of the artificial intelligence-enabled electrocardiography (AI-ECG) model in detecting left ventricular dysfunction, defined as left ventricular ejection fraction (LVEF) ≤ 40% as confirmed by transthoracic echocardiography.

CONTACTS AND LOCATIONS:
Locations (13):
- Taiwan (13):
  - Hualien Armed Forces General Hospital, Hualien City
  - Kaohsiung Armed Forces General Hospital Gangshan Branch, Kaohsiung City
  - Kaohsiung Armed Forces General Hospital, Kaohsiung City
  - Zuoying Armed Forces General Hospital, Kaohsiung City
  - Tri-Service General Hospital Keelung Branch, Keelung
  - Tri-Service General Hospital Penghu Branch, Pengfu
  - Kaohsiung Armed Forces General Hospital Pingtung Branch, Pingtung City
  - Taichung Armed Forces General Hospital Zhongqing Branch, Taichung
  - Taichung Armed Forces General Hospital, Taichung
  - Tri-Service General Hospital Beitou Branch, Taipei
  - Tri-Service General Hospital Songshan Branch, Taipei
  - Taoyuan Armed Forces General Hospital Hsinchu Branch, Taoyuan District
  - Taoyuan Armed Forces General Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen HY, Lin CS, Fang WH, Lou YS, Cheng CC, Lee CC, Lin C. Artificial Intelligence-Enabled Electrocardiography Predicts Left Ventricular Dysfunction and Future Cardiovascular Outcomes: A Retrospective Analysis. J Pers Med. 2022 Mar 13;12(3):455. doi: 10.3390/jpm12030455. PMID 35330455